CLINICAL TRIAL: NCT03434106
Title: Sjögren's Syndrome Is Associated With Meibomian Gland Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: LanZhou University (Other)
Responsible Party: Principal Investigator, Jingmin Yuan, MD, MD, LanZhou University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018A-005
Record Dates: First submitted 2018-02-09; First posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Meibomian Gland Dysfunction; Sjögren's Syndrome
Keywords: meibomian gland dysfunction; Sjögren's syndrome; dry eye disease
MeSH Terms: conditions — Meibomian Gland Dysfunction; Sjogren's Syndrome; Dry Eye Syndromes | interventions — carbomer; Dextrans

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- primary Sjögren's syndrome (Experimental): The female patients with primary Sjögren's syndrome receive the Tears Naturale Forte and Liposic.
  Interventions: Drug: liposic; Drug: Tears Naturale Forte
- secondary Sjögren's syndrome (Experimental): The female patients with secondary Sjögren's syndrome receive Tears Naturale Forte and Liposic.
  Interventions: Drug: liposic; Drug: Tears Naturale Forte
- meibomian gland dysfunction (Experimental): The female patients with meibomian gland dysfunction receive the Tears Naturale Forte and Liposic.
  Interventions: Drug: liposic; Drug: Tears Naturale Forte
- control (Experimental): the female had no history of autoimmune disease receive the Tears Naturale Forte and Liposic.
  Interventions: Drug: liposic; Drug: Tears Naturale Forte

INTERVENTIONS:
Drug: liposic — Liposic eye gel contain the active ingredient carbomer, which is a type of medicine known as an eye lubricant. It is used for the treatmen
  Other Names: Carbomer
Drug: Tears Naturale Forte — This medication is used to relieve dry, irritated eyes
  Other Names: DEXTRAN/HYPROMELLOSE/GLYCERIN

SUMMARY:
The investigators hypothesize that the dry eye caused by SS may include the evaporative type, resulting from the MGD. Furthermore, the investigators hypothesize that both pSS and sSS are associated with MGD.To test our hypothesis, we conducted a prospective clinical study in patients with SS (both pSS and sSS) and MGD, and the normal population All subjects were matched for both age and gender and assessed for tear function and ocular surface signs and symptoms.

ELIGIBILITY:
Inclusion Criteria:

* All the subjects are female and age between 50-60 years
* Patients with primary SS fulfilled the criteria established by the European Study Group
* Patients with SLE and RA met the criteria set by the American College of Rheumatology

Exclusion Criteria:

* The control history of autoimmune disease

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-02-10 (Actual); Primary Completion 2018-05-31 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Ocular Surface Disease Index | up to 3 months after tear substitutes apply
  The OSDI questionnaire is used to quantify the dry eye symptoms. Subjects will be asked questions regarding the dry eye symptoms that they had experienced; the OSDI questions is drawn from 3 different subscales: ocular symptoms, vision-related functions, and environmental triggers. Each answer is scored on a 4-point scale from zero (indicating no problems) to four (indicating a significant problem). Responses to all of the questions are combined to generate a composite OSDI score that ranges from 0 to 100, with higher OSDI scores indicating more severe symptoms. Symptoms of dry eye, such as dryness, burning, foreign body sensation, stabbing pain, photophobia, and visual fluctuations, are also noted
meibomian gland function | up to 3 months after tear substitutes apply
  assessment of the quality of meibomian gland secretions, according to a published classification system (21). In brief, the grading scheme was "0" for clear excreta with small particles, "1" for opaque excreta with normal viscosity, "2" for opaque excreta with increased viscosity, and "3" for secreta that retained shape after digital expression.
fluorescein staining of the cornea | up to 3 months after tear substitutes apply
  Upper, lower, nasal, temporal and central quadrants were used. Superficial punctate keratopathy (SPK) in the cornea was scored from 0 to 3 in each quadrant: 0, no staining in the cornea; 1, <5 punctuate stains; 2, >5 punctuate stains but <10; and 3, >10 or filamentous staining detected. The total number was obtained by adding the scores of the four quadrants for each eye (0-15).
noninvasive tear breakup time | up to 3 months after tear substitutes apply
  Four IR diodes were set on the Keratograph 5 (Oculus, Wetzlar, Germany) and arranged in two pairs, located one above the other. The red ring illumination used for corneal topography was deactivated; this ensured a dark background for the examination. An illuminated ring pattern was then projected onto the cornea. At the start of the recording, the subject will be asked to blink his or her eyes three times and then to keep them open as long as possible. Irregularities in the reflected image will be observed closely. Special attention will be given to distortions and gaps in individual rings and the time such deviations from the original ring pattern took to occur. The examination will be recorded on video.
Schirmer's test with and without anesthesia | up to 3 months after tear substitutes apply
  The Schirmer test without anesthesia (S1T) for tear secretion function will be performed by inserting a 30-mm Schirmer tear test strip (Jingming, Tianjing, China) into the inferior fornix at the junction of the middle and lateral thirds of the lower eyelid margin. Schirmer test strips will remain in place for 5 minutes with the eyes closed. The extent of wetting will be subsequently measured according to the scale provided by the manufacturer. Potential scores ranged from 0 to 30 mm, with lower scores indicating greater tear production abnormalities.

SECONDARY OUTCOMES:
tear meniscus | up to 3 months after tear substitutes apply
  The subject will be asked to blink her eyes once ,then the image of tear meniscus height will be captured by a Keratograph 5 (Oculus, Wetzlar, Germany).After that tear meniscus height will be measured at the centre of the lower lid margin. This performance will be taken three times and the average value will be recorded.
rose bengal staining of the conjunctiva | up to 3 months after tear substitutes apply
  rose bengal staining (graded on a 0-3 scale) of the conjunctiva (six nasal and temporal areas) and the whole cornea.

CONTACTS AND LOCATIONS:
Locations (1):
- Lanzhou University Second Hospital, Lanzhou, Gansu, China